CLINICAL TRIAL: NCT05284396
Title: Involved Nodal Irradiation vs Involved Field Irradiation After Cth in Ttt of Early Stages HDs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Esam Eldin Hassan, Marwa Esam Eldin, Assiut University
Other Study IDs: radiotherapy in lymphomas
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: IFRT vs NFRT — involved field irradiation versus nodal field irradiation

SUMMARY:
determine the early toxicity and loco-regional control comparing outcome of radiothrapy rither by using INRT or IFRT in treatment of early stage hodgkin lymphoma

determine progression-free survival and late toxisty

DETAILED DESCRIPTION:
Hodgkin lymphoma (HL) is one of the most frequent lymphomas in the Western world, with an annual incidence of about 3 cases per 100,000 persons. This lymphoid malignancy involves peripheral lymph nodes and can also affect organs such as liver, lung, and bone marrow. About 40% of patients suffer from constitutional symptoms ("B-symptoms"). Based on differences in the histological picture and the phenotype of the tumor cells, HL is subclassified into nodular sclerosis, mixed cellularity, lymphocyte-rich, lymphocyte-depleted, and nodular lymphocyte-predominant HL (NLPHL) (1) Hodgkin lymphoma is estimated to account for about 10% of cases of newly diagnosed lymphoma in the United States (8,260 of 80,500), the remainder being Non-Hodgkin lymphoma. Of 21,210 estimated deaths yearly due to lymphoma, about 1,070 (or 5%) are from Hodgkin lymphoma. It accounts for about 0.5% of newly diagnosed cases of cancer in the United States and about 0.2% of all cancer deaths. However lymphoma is the most common cancer diagnosed in adolescents (aged 15 to 19 years) accounting for 21% of new diagnoses, almost two-thirds of which is Hodgkin lymphoma (2) In patients with Hodgkin lymphoma, a definitive diagnosis is critical and requires that the treating physician provide the pathologist with an adequate pathologic specimen. Fine-needle aspiration or core-needle biopsy specimens are commonly inadequate because they do not represent the architecture of the lymph node and therefore preclude an accurate diagnosis. Hodgkin lymphoma has the unique characteristic of malignant cells constituting only a minority of the intratumoral cell population, and therefore, a small biopsy specimen may not include sufficient malignant cells.(3)

To establish a definitive diagnosis, it is necessary to identify Reed-Sternberg cells within the biopsy specimen. These cells are commonly seen within a rich cellular environment composed of reactive lymphocytes, eosinophils, and histiocytes. Two distinct disease entities have been defined in Hodgkin lymphoma, the commonly diagnosed classical Hodgkin lymphoma and the uncommon nodular lymphocyte-predominant Hodgkin lymphoma.(4)

The past few decades have seen significant progress in the management of pt with HL, it is curable in at least 80% of patient. Early stage Hodgkin's lymphoma (HL) patients treated with a combination of chemotherapy and radiotherapy have an excellent clinical outcome, with overall survival of approximately 90% [5].

With modern techniques, including better CT scan imaging, FDG-PET/CT scans and more accurate radiation technology ,It is now possible to customize radiotherapy for each patient with accurate delivery of radiation to the initially involved volume while minimizing the radiation dose to normal tissues(6).

The advent of combined modality treatment had previously led to a Shift in practice from extended field radiotherapy techniques to involved Field radiotherapy (IFRT)(7-8).

Some recent studies have shown the safety of further reductions in field sites. With the concept of involved node radiotherapy (INRT) in order to reduce the risk of radiotherapy-induced toxicity. INRT is based on treating only initially involved lymph nodes and excluding adjacent uninvolved nodal areas(9-11)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven Hodgkin's Lymphoma, with exclusion of the nodular lymphocyte predominant subtybe
* Clinical stage I or II, only supra-diaphragmatic nodes, both favorable and unfavorable prognostic subsets
* Previously untreated.
* Age: between 18 and 75 years.
* Good general condition(WHO performance status 0-2).
* Free of concurrent disease.

Exclusion Criteria:

* Patients with impaired heart, lung, liver, or kidney function.
* Previous malignant diseases or HIV-positive status
* Patient with advanced or infra-diaghragmatic Hodgkin's disease
* Pregnant or lactating women
* Patient with prior irradiation to the neck and thorathic region

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: statistical analyses were performed using IBM SPSS Statistics version 20 (SPSS Inc., Chicago, IL, USA). Categorical data were presented as frequencies and percentages, while Chi-square test was used for comparisons between groups. Continuous data were reported as means ±standard deviations and students' T-test was used for comparisons between groups. For comparison between progression free survival ,Kaplan-Mayar survival curve and log-rank test were performed. In all statistical tests p-value <0.05 was considered statistically significant.
  •Sample size: All pt who met at inclusion criteria at SECI will be included in our study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between different irradiation modalities in tretment of early stage hodgkin lymphoma | baseline
  involved nodal Irradiation versus Involved field Irradiation after Chemotherapy in treatment of Early stage Hodgkin's lymphoma